CLINICAL TRIAL: NCT00812708
Title: Clinical Evaluation of Morcher Artificial Iris Diaphragms to Treat Light and Glare Sensitivity in Partial or Complete Aniridia
Brief Title: Clinical Evaluation of Morcher Artificial Iris Diaphragms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Kevin M. Miller, MD, Kolokotrones Chair in Ophthalmology, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-06-072
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Aniridia; Iris; Deformity
Keywords: aniridia; Morcher iris diaphragms; modified capsule tension ring; artificial iris; iris reconstruction lens; glare sensitivity; photophobia
MeSH Terms: conditions — Aniridia; Congenital Abnormalities; Photophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Morcher iris diaphragm implantation (Experimental): This is a non-randomized, non-comparative interventional surgical series. Patients will undergo Morcher iris diaphragm implantation in their affected eye(s). After surgery, patients will complete 5 postoperative examinations. At each examination, they will be evaluated for changes in light and glare sensitivity and visual acuity. They will also be monitored for adverse reactions.
  Interventions: Device: Morcher iris diaphragm implantation

INTERVENTIONS:
Device: Morcher iris diaphragm implantation — Surgical implantation of Morcher iris device(s)
  Other Names: Morcher device models: 96F, 96S, 50D, 50F, and 67B

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Morcher iris diaphragms in the treatment of congenital and acquired aniridia. Morcher iris diaphragms are intraocular devices that are designed to provide an artificial pupil for patients suffering from partial or complete aniridia. These devices are constructed from clinical quality, ultraviolet light-absorbing, opaque black polymethylmethacrylate (PMMA). After surgical implantation, patients are monitored over the course of 1 year to measure any changes to visual acuity and improvements in light and glare sensitivity.

DETAILED DESCRIPTION:
Aniridia is a condition in which the iris, the colored portion of the eye, is either partially or completely absent. The iris is responsible for regulating the amount of light entering the eye by adjusting the size of the pupil.

Aniridia can either be a congenital condition, often a genetically-based abnormality affecting the formation of the iris, or it can be acquired by blunt trauma with or without rupture, penetrating trauma, or severe intraocular inflammation.

Aniridia can also vary in the level of severity. A mild case might involve a thinner iris or iris remnant with a normal pupil. A severe case might involve complete absence of the iris or impairment of the muscles responsible for adjusting pupil size.

Iris defects can occur without the loss of stromal tissue as well. In some cases, the iris pigment epithelium is missing. In other cases, holes are present in the iris or the pupil is chronically enlarged or mydriatic.

People who suffer from iris defects also commonly suffer from other eye conditions. Common comorbidities include glaucoma, cataract, and nystagmus. Other structures in the eye are often affected, including the cornea, crystalline lens, zonules, and retina. Iris defects can cause severe visual disability if untreated.

Common treatments for iris defects include the use of colored or tinted glasses or contact lenses to reduce the amount of light entering the eye.

In this trial, several Morcher iris diaphragms are being evaluated as a potential treatment to improve the symptoms associated with aniridia and other iris defects. Morcher iris diaphragms are manufactured in Germany by Morcher GmbH [website: http:// www.morcher.com]. These devices have been utilized in Europe to treat aniridic patients for over 40 years. Additionally, these devices hold the European CE mark of conformity.

When a patient is implanted with a Morcher iris device, surgery always involves additional standard of care surgical procedures. Typically, a device is implanted during cataract surgery along with an intraocular lens (IOL). Morcher devices can also be implanted during an IOL exchange with or without an anterior vitrectomy. All implantation procedures take place in an operating room under local or general anesthesia. In some cases, a Morcher iris reconstruction lens containing both an artificial iris and a lens is implanted. Also, depending on the condition of the eye, the lens and iris device may need to be sutured to the sclera, the white portion of the eye.

All patients undergoing surgery are prescribed 2 different eye drops, an antibiotic and a corticosteroid. These medications are used for up to 6 weeks following implantation of the device. There are 5 postoperative follow-up visits that each patient must complete. Visits occur at specific intervals over the course of a 1-year period. At each visit, standard of care procedures are performed and, at certain time points during the follow-up interval, digital photos and endothelial cell counts are obtained. In instances where both eyes are implanted, surgery for the second eye is scheduled 6 months or more later.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years old and have partial or complete aniridia.
* Be willing and able to comply with all follow-up requirements.
* Must have increased light and/or glare sensitivity or complete aniridia.
* Patients may be phakic, aphakic, or pseudophakic.
* Phakic patients will require simultaneous cataract surgery.
* Aphakic patients will require secondary intraocular lens implantation.

Exclusion Criteria:

* The presence of any ocular condition that may cause complications from the surgical procedure
* Active ocular infection or inflammation
* Patients with allergies to operative and/or postoperative medications
* Pregnant or lactating women
* Persons who, in the determination of the investigator, are not competent to understand the procedure or the actions asked of them as research subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-04-09 (Actual); Primary Completion 2014-06-20 (Actual); Study Completion 2021-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Miller, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Stein Eye Institute, UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung MY, Miller KM, Weissman BA. Morcher iris reconstruction lens and rigid contact lens for traumatic aniridia. Eye Contact Lens. 2009 Mar;35(2):108-10. doi: 10.1097/ICL.0b013e318199b00b. PMID 19265334
- [Result] Olson MD, Masket S, Miller KM. Interim results of a compassionate-use clinical trial of Morcher iris diaphragm implantation: report 1. J Cataract Refract Surg. 2008 Oct;34(10):1674-80. doi: 10.1016/j.jcrs.2008.05.048. PMID 18812117
- [Result] Date RC, Olson MD, Shah M, Masket S, Miller KM. Outcomes of a modified capsular tension ring with a single black occluder paddle for eyes with congenital and acquired iris defects: Report 2. J Cataract Refract Surg. 2015 Sep;41(9):1934-44. doi: 10.1016/j.jcrs.2015.10.001. PMID 26603402
- [Result] Miller KM, Nicoli CM, Olson MD, Shah M, Masket S. Outcomes of implantation of modified capsule tension rings with multiple black occluder paddles for eyes with congenital and acquired iris defects: Report 3. J Cataract Refract Surg. 2016 Jun;42(6):870-8. doi: 10.1016/j.jcrs.2016.03.035. PMID 27373394
- [Result] Lin SR, Miller KM. Lessons Learned from Implantation of Morcher 50D and 96S Artificial Iris Diaphragms. Case Rep Ophthalmol. 2017 Nov 23;8(3):527-534. doi: 10.1159/000484128. eCollection 2017 Sep-Dec. PMID 29515428
- [Result] Miller KM, Kuo A, Olson MD, Masket S. Safety and efficacy of black iris diaphragm intraocular lens implantation in eyes with large iris defects: Report 4. J Cataract Refract Surg. 2018 Jun;44(6):686-700. doi: 10.1016/j.jcrs.2018.03.033. Epub 2018 Jul 4. PMID 30041739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Most patients were recruited from the principal investigator's ophthalmic practice. A few were referred by local ophthalmologists.
Groups:
- Morcher Iris Diaphragm Study Group: This group consists of all patients enrolled in the Morcher iris diaphragm study.
Period: Overall Study
Arm/Group | Morcher Iris Diaphragm Study Group
Started | 72 (6 patients withdrew from the study before being taken to the operating room.)
Taken to Surgery for Device Implantation | 66 (2 patients could not be implanted because of intraoperative complications.)
Completed | 64
Not Completed | 8
Not completed — Device could not be implanted | 2
Not completed — Lack of medical insurance | 1
Not completed — Switched to another study | 1
Not completed — Surgery cancelled due to uveitis | 1
Not completed — Signed consent but later withdrew | 3

BASELINE CHARACTERISTICS:
Population: One eye per patient was enrolled, thus the number of study eyes equals the number of study participants.
Groups:
- Morcher Iris Diaphragm Study Group: Seventy two patients signed consent forms to participate in the Morcher iris diaphragm study.
Arm/Group | Morcher Iris Diaphragm Study Group
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 47
  More than one race | 0
  Unknown or Not Reported | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Change in Light and Glare Sensitivity as Determined by a Clinical Glare Test (Primary Efficacy Measure)
Description: The primary efficacy measure of the study was the change in corrected distance visual acuity (CDVA) under glare conditions. A transilluminator light was held just in front of the distance corrected study eye in one of four quadrants (above, below, nasal, or temporal) to the line of sight to evoke a glare response. The direction that produced the worst CDVA was called the CDVA with glare. A ≥ 2 line improvement in Snellen CDVA with glare following Morcher device implantation was considered a positive clinical change (glare sensitivity better). A ≥ 2 line worsening of Snellen CDVA with glare following Morcher device implantation was considered a negative clinical change (glare sensitivity worse). A change of < 2 Snellen lines following Morcher device implantation was considered to be a neutral change (glare sensitivity the same).
Time Frame: Preoperatively and 1 year postoperatively
Population: This group consisted of all patients implanted with Morcher iris diaphragms.
Measure: Count of Participants; unit: Participants
Groups:
- Morcher Iris Diaphragm Implantation Group: All patients implanted with Morcher iris diaphragms.
Arm/Group | Morcher Iris Diaphragm Implantation Group
Number analyzed (Participants) | 64
Participants
  Glare sensitivity better | 51
  Glare sensitivity the same | 12
  Glare sensitivity worse | 1

2. Primary Outcome: Change in Best Corrected Visual Acuity (Primary Safety Measure)
Description: The primary safety measure of the study was the change in best corrected distance visual acuity (CDVA) as measured using a Snellen eye chart. A ≥ 2 line improvement in Snellen CDVA following Morcher device implantation was considered a positive clinical change (visual acuity better). A ≥ 2 line worsening of Snellen CDVA following Morcher device implantation was considered a negative clinical change (visual acuity worse). A change of < 2 lines was considered to be a neutral change (visual acuity the same).
Time Frame: Preoperatively and 1 year postoperatively
Population: This group consisted of all patients implanted with Morcher iris diaphragms.
Measure: Count of Participants; unit: Participants
Arm/Group | Morcher Iris Diaphragm Implantation Group
Number analyzed (Participants) | 64
Participants
  Visual acuity better | 35
  Visual acuity the same | 28
  Visual acuity worse | 1

3. Secondary Outcome: Change in Glare Sensitivity Under Day Time Lighting Conditions (Secondary Efficacy Measure)
Description: A secondary efficacy measure of the study was day time glare disability as assessed by subjective questionnaire. Glare disability was rated using a 0 to 10 scale, where 0 was considered very slight and 10 was considered very significant.
Time Frame: Preoperatively and 3 months postoperatively
Population: This group consisted of all patients implanted with Morcher iris diaphragms.
Measure: Count of Participants; unit: Participants
Groups:
- Morcher Iris Diaphragm Implantation Group: Glare sensitivity was assessed by a questionnaire that was scored on a 0 to 10 scale under daytime and nighttime lighting conditions.
Arm/Group | Morcher Iris Diaphragm Implantation Group
Number analyzed (Participants) | 64
Participants
  Subjective day time glare sensitivity better | 57
  Subjective day time glare sensitivity the same | 5
  Subjective day time glare sensitivity worse | 2

4. Secondary Outcome: Change in Glare Sensitivity Under Night Time Lighting Conditions (Secondary Efficacy Measure)
Description: Another secondary efficacy measure of the study was night time glare disability as assessed by subjective questionnaire. Glare disability was rated using a 0 to 10 scale, where 0 was considered very slight and 10 was considered very significant.
Time Frame: Preoperatively and 3 months postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Morcher Iris Diaphragm Implantation Group
Number analyzed (Participants) | 64
Participants
  Subjective night time glare sensitivity better | 56
  Subjective night time glare sensitivity the same | 5
  Subjective night time glare sensitivity worse | 3

5. Secondary Outcome: Change in Endothelial Cell Count (Secondary Safety Measure)
Description: A secondary safety measure of the study was the change in endothelial cell count. A loss of >10% of central corneal endothelial cells was considered clinically significant at the onset of the study. (Note, the 10% loss criterion was established before the 67B implant was added to the list of study devices. The 67B implant has an expected greater cell loss than that associated with the 96F, 96S, 50D, and 50F modified capsule tension rings because it requires a larger incision for implantation. Thirty one (48.4%) of the 64 patients were implanted with the 67B device.)
Time Frame: Preoperatively and 3 months postoperatively
Population: This group consisted of all patients implanted with Morcher iris diaphragms, for whom simultaneous corneal transplantation was not performed, and in whom endothelial cell counts could be obtained preoperatively and postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Morcher Iris Diaphragm Implantation Group
Number analyzed (Participants) | 35
Participants
  Endothelial cell loss ≤ 10% | 17
  Endothelial cell loss > 10% | 18

6. Secondary Outcome: Need to Explant or Exchange a Morcher Iris Diaphragm (Secondary Safety Measure)
Description: Another secondary safety measure of the study was the need to explant or exchange a Morcher iris diaphragm within 1 year of implantation. Explantation in < 25% of patients was considered to be clinically acceptable.
Time Frame: Preoperatively and 1 year postoperatively
Population: This group consisted of all patients implanted with Morcher iris diaphragms.
Measure: Count of Participants; unit: Participants
Arm/Group | Morcher Iris Diaphragm Implantation Group
Number analyzed (Participants) | 64
Participants
  Morcher device explanted | 1
  Morcher device not explanted | 63

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 year following Morcher iris diaphragm implantation.
Description: Adverse Event and Serious Adverse Event data were collected according to institutional review board (IRB) guidelines.
Arm/Group | Morcher Iris Diaphragm Implantation Group
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 6/64
Other Adverse Events (participants affected / at risk) | 5/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morcher Iris Diaphragm Implantation Group (N=64)
Decentered piggyback intraocular lens (Eye disorders) | 1 (1)
Retained lens fragment (Eye disorders) | 1 (1)
Corneal failure (Eye disorders) | 1 (1)
Corneal graft-host interface leak (Eye disorders) | 1 (1)
Morcher iris diaphragm rotation (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morcher Iris Diaphragm Implantation Group (N=64)
Intraoperative hyphema (Eye disorders) | 1 (1)
Cystoid macular edema (Eye disorders) | 1 (1)
Acute iritis (Eye disorders) | 1 (1)
Ocular hypertension (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No